CLINICAL TRIAL: NCT07313176
Title: A Prospective, Non-Interventional Study on the Long-term Effectiveness of Levodopa-Entacapone-Carbidopa Intestinal Gel (LECIGON®) in Patients With Parkinson's Disease Previously Treated With Subcutaneous Foslevodopa in Routine Care
Brief Title: Long Term Effectiveness of Levodopa-Entacapone-Carbidopa Intestinal Gel in Participants With Advanced Parkinson's Disease
Acronym: SWITCH-ON
Status: Recruiting | Type: Observational
Sponsor: Britannia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-MA-2025-01
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Parkinson Disease
Keywords: Parkinson´s Disease; Movement Disorders; Portable Pump; Neurodegenerative Disorder; Subcutaneous Foslevodopa; Quality of Life; Dopamine Agonists
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Receiving LECIGON® Treatment: All participants with advanced Parkinson's disease who switched from subcutaneous foslevodopa (foslevodopa-foscarbidopa) to LECIGON®, will be observed in the study. Participants real-world data on the long-term effectiveness of LECIGON® in routine clinical practice will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary objective of the study is to assess the effectiveness of LECIGON® treatment on the reduction in OFF time (h/day) from baseline at 12 months as measured by Movement Disorder Society-Unified Parkinson's Disease Rating Scale, Part IV (MDS-UPDRS IV).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18 years old and over) with advanced Parkinson's disease with severe motor fluctuations and dyskinesia
* Participants for whom the treating physician has made the decision to initiate treatment with LECIGON® in accordance with the Summary of Product Characteristics (SmPC)
* Participants must have had previous treatment with subcutaneous foslevodopa (foslevodopa-foscarbidopa) for a minimum of 1 month
* Participants or legal representative must have signed informed consent to participate in the study

Exclusion Criteria:

* Participants with contraindications as defined in the current version of the SmPC for LECIGON®
* Participants who will not be seen again for their follow up care at the investigator's site after commencement of LECIGON® therapy
* Participants with anticipated pump placement or pump use issues, e.g. participants with acute severe illness, participants unable to perform pump therapy, and in case of lacking compliance due to severe dementia, agitation or alcohol abuse
* Participants taking part in a clinical (interventional) trial at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with advanced Parkinson's disease have discontinued treatment with foslevodopa-foscarbidopa and are receiving LECIGON® as part of their routine care will be included in this observational study.
Sampling Method: Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Reduction in OFF time (h/day) as Measured by Movement Disorder Society-unified Parkinson's Disease Rating Scale, Part IV (MDS-UPDRS IV) at 12 months | Baseline, Month 12
  The MDS-UPDRS is a revision of the Unified Parkinson's disease rating scale (UPDRS) developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part IV concerns motor complication and all questions in Part IV that deal with motor fluctuations and dyskinesias, the investigator is required to conduct the interview of participants.

SECONDARY OUTCOMES:
Change from Baseline in the Reduction in OFF time (h/day) as Measured by MDS-UPDRS IV at 6 months | Baseline, Month 6
  The MDS-UPDRS is a revision of the UPDRS developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part IV concerns motor complication and all questions in Part IV that deal with motor fluctuations and dyskinesias, the investigator is required to conduct the interview of participants.
Change from Baseline in the Reduction in OFF time (h/day) as Measured by Hauser Patient Diaries | Baseline, Months 6 and 12
  The Hauser Diary is a home diary, completed by the participant, that assesses functional status in participants with Parkinson's disease with motor fluctuations and dyskinesia. Participants will complete the Hauser Diary for a 72-hour period occurring after informed consent has been obtained and prior to LECIGON® treatment start and for 48 hours prior to each of the two follow-up visits.
Change from Baseline in LECIGON® Treatment Patterns due to Change in Daily Levodopa Dose (mg/day) as Measured by Total Daily Dose Using Multi-rate Programming of Pump | Baseline, Months 6 and 12
  Total daily levodopa dose will be measured using the multi-rate programming of pump.
Change from Baseline in Clinical Global Impression of Improvement as Measured by Clinical Global Impression of Change (CGI-C) | Baseline, Months 6 and 12
Change from Baseline in Clinical Global Impression of Improvement as Measured by Patient Global Impression of Change (PGI-C) at 12 months | Baseline, Months 6 and 12
Change from Baseline in Non-motor Experiences of Daily Living as Measured by MDS-UPDRS-I | Baseline, Months 6 and 12
  The MDS-UPDRS is a revision of the UPDRS developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part I concerns non-motor experiences of daily living. Several questions from Part I are designed to be amenable to a patient/caregiver questionnaire format and therefore can be completed without the investigator's input. For the remaining Part I questions that deal with complex behaviors, the investigator is required to conduct the interview of participants.
Change from Baseline in Motor Complications as Measured by MDS-UPDRS-IV | Baseline, Months 6 and 12
  The MDS-UPDRS is a revision of the UPDRS developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part IV concerns motor complication and all questions in Part IV that deal with motor fluctuations and dyskinesias, the investigator is required to conduct the interview of participants.
Change from Baseline in Quality of Life as Measured by Parkinson's Disease Questionnaire Total Score (PDQ-8) | Baseline, Months 6 and 12
  The PDQ-8 is an eight-question instrument, completed by the participants, that measures the quality of life among Parkinson's disease participants. It is a shortened version of the 39-item Parkinson's disease questionnaire to reduce participant burden and increase convenience for use among Parkinson's disease participants. It includes one question from each of the dimensions including include mobility, activities of daily of living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.
Change from Baseline in Sleep as Measured by Parkinson's Disease Sleep Scale - 2 (PDSS-2) | Baseline, Months 6 and 12
  The PDSS is a visual analogue scale, completed by the Parkinson's disease participant, addressing 15 commonly reported symptoms associated with sleep disturbances, including overall quality of night's sleep, sleep onset and maintenance insomnia, nocturnal restlessness, nocturnal psychosis, nocturia, nocturnal motor symptoms, sleep refreshment, and daytime dozing. The PDSS-2 uses a 5-point frequency scale (0-4) for each item, with a total score ranging from 0 to 60. Higher scores indicate more severe sleep problems.
Treatment Satisfaction Questionnaire at Months 6 and 12 | At Months 6 and 12
  Participants will be asked questions to assess their satisfaction with LECIGON® treatment.
Change from Baseline in Body Mass Index (BMI) | Baseline, Months 6 and 12
Number of Participants With Adverse Drug Reactions (ADRs), Serious ADRs, Reportable Events (REs), Serious REs and REs of Special Interest (RESIs) | 12 months
  An ADR is any untoward and unintended response to a medicinal product, related to any dose administered and which implies a RE with at least a reasonable possibility of a causal relationship with the use of the product. A RE is any unfavorable or unintended sign, symptom or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. RESIs include drug interaction, drug exposure during pregnancy, drug exposure during breastfeeding, lack of drug efficacy, overdose, misuse/abuse, medication errors (incl. prescription and application errors), off-label use, adverse reaction which occurred during occupational exposure, falsified medicinal product, suspected transmission of infectious agents via a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Amlani, MPharm, Study Director — Britannia Pharmacetuicals
Locations (2):
- Spain (2):
  - Virgen del Rocío University Hospital, Seville, Av. Manuel Siurot, S/n
  - Complejo Hospitalario Universitario de A Coruña (CHUAC), A Coruña

IPD SHARING:
Plan to Share IPD: No